CLINICAL TRIAL: NCT04351854
Title: Registry for Clinical Presentation and Management of Patients With COVID-19 in the Emergency Room
Acronym: ReCovER
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr. med., University of Cologne
Other Study IDs: ReCovER
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Corona Virus Infection; SARS-CoV 2
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SARS-CoV-2-infection: Patients with clinical suspicion or evidence of SARS-CoV-2-infection on presentation in the ED
  Interventions: Other: Retrospective data collection
- Control group: Particularly, controls will be identified retrospectively at the same hospitals based on matching of demographics, underlying diseases and duration of hospital stay (i.e. one control per case, both in the same hospital). Moreover, the mere suspicion of SARS-CoV-2-infection on admission in the ED is sufficient for enrolment. A considerable portion of these patients are actually not infected and serve as internal control.
  Interventions: Other: Retrospective data collection

INTERVENTIONS:
Other: Retrospective data collection — Retrospective data collection to identify predicting factors in the clinical picture of COVID-19 patients presenting to the ED.

SUMMARY:
Patients with COVID-19 usually present in the ED and receive their initial medical check-up here. We will try to gather information of comorbidities and other conditions at the time of presentation of COVID-19 patients to the ED. The course of the disease prior to admission as well as the momentary health status at presentation to the ED are of interest because they influence risk stratification and decision-making of treating physicians. The ratio of patients with mild or moderate to severe symptoms will help to calculate the need for hospital beds including beds on Intensive Care Units (ICU) and Intermediate Care Units (IMC), as well as the need for other hospital resources.

DETAILED DESCRIPTION:
Patients with COVID-19 usually present in the ED and receive their initial medical check-up here. It is the ED where crucial diagnostic and therapeutic steps are taken and where the decision for admission or discharge is made. As of now, the effectiveness and value of these initial measures and decisions are unclear. With still raising numbers of infections despite regulatory constraints in place, there is an urgent need to develop valid decision trees on how to treat patients suspected with COVID-19 in the ED.

Apart from the already described risk factors little is known about if and to which degree an infection with COVID-19 itself predisposes to other acute conditions (e.g. myocarditis, myocardial infarction or stroke). We will try to gather information of comorbidities and other conditions at the time of presentation of COVID-19 patients to the ED.

Not all patients seek medical consultation at the very beginning of symptoms. The course of the disease prior to admission as well as the momentary health status at presentation to the ED are of interest because they influence risk stratification and decision-making of treating physicians. For example: an immunocompromised patient who presents with mild symptoms at a very early stage of COVID-19 would probably be deemed more at risk than the same patient who reports mild symptoms without progression for a duration of several weeks.

The ratio of patients with mild or moderate to severe symptoms will help to calculate the need for hospital beds including beds on Intensive Care Units (ICU) and Intermediate Care Units (IMC), as well as the need for other hospital resources. It will also help to identify the need for capacities in ambulatory care. COVID-19 Patients with mild or moderate symptoms can remain in quarantine at home. This would not only disburden hospitals but would also lower the risk for previously uninfected patients otherwise having to share rooms and wards with them.

Confirming the diagnosis There is uncertainty with regard to the best initial diagnostic in COVID-19 patients. Diagnostic tool of choice is a low-dose CT-scan of the thorax, which will detect typical radiologic signs of COVID-19 (ground-glass-opacities, bilateral consolidations and "crazy paving") with a high sensitivity, and in some cases even before onset of clinical symptoms. However, these features are also seen in other viral pneumonias and specificity reaches only 25%. Moreover, a CT-scan might not be available 24/7 in all hospitals, is time-consuming and exposes radiologic personnel to the risk of infection. Additionally, as is described later, many patients present with severe hypoxemia, a situation in which they might not be able to lie in a supine position in the CT-scanner. The role of lung ultrasound (LUS) in detection of COVID-19 has not been examined properly so far.

Testing for COVID-19 usually is done using an oral swab (or expectorated sputum) and real-time PCR (RT-PCR) after a clinical suspicion based on different parameters and/or after visits of the patient to regions with high prevalence of SARS-CoV-2. The sensitivity of this method has not been systematically evaluated, however, false-positive, as well as false-negative results have been reported. Moreover, there are sometimes contradictory results of RT-PCR and CT-scan. The registry will be used to collect and compare diagnostic data from radiological exams as well as RT-PCR-testing.

Many COVID-19 patients present with shortness of breath and hypoxemia. Physicians have used different therapeutic approaches including high-flow oxygen (HFNC), non-invasive ventilation or intubation and mechanical ventilation. While a trial with non-invasive methods is deemed safe and adequate by most experts, others have raised concerns and advocate early intubation and invasive ventilation in COVID-19. Participants of the registry will be asked to state the method of oxygenation/ventilatory support that was initiated in the ED.

Admission vs. discharge As has already been laid out, patients with COVID-19 exhibit symptoms of different severity. It is neither possible nor would it be reasonable to hospitalize every patient in which the condition is suspected or confirmed. Unfortunately, there are no diagnostic markers or laboratory cut-offs that help decide if a COVID-19 patient who presents to the ED has to be hospitalized or can be safely managed in ambulatory care. Our goal is to gather information of outcomes in both hospitalized and discharged patients and to compare this data with epidemiological, clinical, laboratory and radiologic data from the date of their visit to the ED.

The ED is the first contact to a hospital. Diagnostic and therapeutic measures from patients who are hospitalized due to the severity of their disease will be analyzed as well as complications or death during hospitalization. The duration of hospitalization will be analyzed and compared to the initial clinical picture.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion or evidence of SARS-CoV-2-infection on presentation in the ED

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical suspicion or evidence of SARS-CoV-2-infection on presentation in the ED and matching controls, based on demographics, underlying diseases and duration of hospital stay (i.e. one control per case, both in the same hospital).
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Identification of risk factors present at the earliest stage of hospital care (i.e. in the ED) that warrant hospital admission. | 6 months
  Identification of risk factors present at the earliest stage of hospital care (i.e. in the ED) that warrant hospital admission.

SECONDARY OUTCOMES:
Determination of the course of the disease (days since onset of symptoms, nature of symptoms, e.g. fever, chills, headache) and the state at which patients present to the ED | 6 months
  Determination of the course of the disease (days since onset of symptoms, nature of symptoms, e.g. fever, chills, headache) and the state at which patients present to the ED
Identification of the ratio of patients with mild or moderate to severe disease | 6 months
  Identification of the ratio of patients with mild or moderate to severe disease

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No